CLINICAL TRIAL: NCT00266383
Title: The Molecular Mechanism and the Role of NRAMP 1gene on Tuberculosis in Taiwan Aboriginal Tribes Population
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Other Study IDs: DOH94-DC-1009
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2005-12-19 (Estimated); Status verified 2005-12

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The human homologue of mice natural-resistance-associated macrophage protein 1 (Nramp 1) gene, NRAMP 1, has been reported to play a role in the susceptibility to tuberculosis in humans. The aboriginal population in Taiwan has a 5-fold higher prevalence of tuberculosis than the Han Chinese. Whether genetic factors such as NRAMP 1 polymorphisms play a role in the prevalence of tuberculosis in Taiwanese aboriginals should be clarified.

ELIGIBILITY:
Inclusion Criteria:

* The NRAMP 1 polymorphism of tuberculous patients in Taiwan.

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250
Dates: Start 2005-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Ih-Jen Su, M.D., Ph.D., Principal Investigator — Division of Clinical Research, National Health Research Institutes
Locations (1):
- National Health Research Institutes, Miaoli County, Taiwan